CLINICAL TRIAL: NCT03481569
Title: Population Pharmacokinetic-pharmacodynamic (PK-PD) Study of 9 Broad-Spectrum Anti-infective Agents in the Cerebro Spinal Fluid (CSF) of Brain Injured Patients With an External Ventricular Drainage (EVD).
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PKpop LCR
Record Dates: First submitted 2018-03-21; First posted 2018-03-29 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Infection
MeSH Terms: conditions — Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Pharmacokinetic study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pharmacokinetic sample (Experimental): Plasma and cerebrospinal fluid samples performed at different timepoint during administration of antibiotic prescribed in routine use
  Interventions: Other: Blood and cerebrospinal fluid pharmacocinetic samples on one of the nine antibiotics prescribed in routine use

INTERVENTIONS:
Other: Blood and cerebrospinal fluid pharmacocinetic samples on one of the nine antibiotics prescribed in routine use — Blood and cerebrospinal fluid pharmacocinetic samples at different time point

SUMMARY:
Nosocomial Central Nervous System infections are difficult to treat and an early appropriate therapy can improve prognosis. The two main reasons for treatments failure are the difficulty to reach high concentrations of antibiotics (ATB) in CNS because of brain barriers (BB), and the emergence of Multi-Drug-Resistant (MDR) pathogens that require high ATB concentrations for being killed. Therefore a better knowledge of ATB CNS distribution and PK-PD characteristics is essential for efficiency of treatments and to avoid resistance progression. Because of BB and cerebrospinal fluid (CSF) turnover, unbound (active) concentrations of ATB in CSF are frequently much lower than corresponding plasma concentrations, which therefore may not be used to predict efficacy. However except for patients with EVD, CSF access is difficult. Overall the litterature about ATB distribution within CSF exist but PK-PD publications are rarer. Especially for Broad Spectrum ATB which are recommended in case of invasive infection in ICU patients due to MDR pathogens such as Acinetobacter baumanii, extended spectrum ß-Lactamase producing (ESBL) pathogens or Multiresistant Staphylococcus aureus.

Furthermore, measuring ATB concentrations within the CSF at certain time-points is necessary but not sufficient to predict antimicrobial efficacy. First PK modelling is required to describe the full CSF concentrations versus time profiles. Then targets must be obtained from literature or determined for the relevant PD index, which may be, depending of the antibiotic, Time over Minimal Inhibitrice Concentration (T>MIC), Area Under the Curve over MIC (AUC/MIC) or peak concentration over MIC (Cmax/MIC). Eventually Monte-Carlo simulations can be conducted to predict the probability of target attainment according to various dosing regimens to find the optimal one.

The goal of this multicenter population PK-PD study is to characterize CSF distribution and challenge recommended dosing regimens of 8 ATB indicated in CNS infections (vancomycin, daptomycin, ceftazidime, meropenem, colistin, linezolid, piperacillin-tazobactam and ceftaroline) and to study the Cefepime diffusion in the CSF, known to be highly neurotoxic.

ELIGIBILITY:
Inclusion Criteria:

* Brain injury patients requiring intensive care management with external ventricular drainage
* Age ≥18 years old
* Patient with a CNS or other site infection treated with one or several of the ATB of the study
* Signed informed consent of the patient or the close friend / family after giving a clear and loyal information about the study
* Free subject, without guardianship or curatorship or subordination
* Patients benefiting from a Social Security system or benefiting from it through a third party

Exclusion Criteria:

* Age under 18 years old
* Acute renal failure defined with a creatinine clearance < 50 mL/min and / or under continuous haemodialysis
* Contraindication to the antibiotic studied
* No informed consent signed or no emergency procedure for continuous infusion antibiotic signed
* Patients not benefiting from a Social Security scheme or not benefiting from it through a third party
* Persons benefiting from enhanced protection, namely minors, persons deprived of their liberty by a judicial or administrative decision, persons staying in a health or social institution, adults under legal protection, and finally patients in emergencies.
* Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2018-07-06 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
CSF-to-plasma area under the unbound concentration-time curve for each antibiotic | 5 days

SECONDARY OUTCOMES:
Time > Minimal Inhibitrice Concentration for each antibiotic | 5 days
Area Under the Curve / Minimal Inhibitrice Concentration for each antibiotic | 5 days
Peak concentration / Minimal Inhibitrice Concentration for each antibiotic | 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHU of Poitiers, Poitiers, France